CLINICAL TRIAL: NCT01970904
Title: A Multicenter, Open-label, Randomized, 3-arm, Phase II Profiling Trial of Pharmacokinetics, Pharmacodynamics and Safety of DEB025/Alisporivir in Combination With Ribavirin Therapy in Chronic Hepatitis C Genotype 2 and 3 Treatment naïve Patients
Brief Title: Pharmacokinetics, Pharmacodynamics and Safety of DEB025 Plus Ribavirin in Chronic Hepatitis C Genotype 2 and 3 Treatment naïve Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDEB025A2222; 2012-004185-17 (EudraCT Number)
Record Dates: First submitted 2013-09-30; First posted 2013-10-28 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C; Liver Disease
Keywords: Chronic hepatitis C; DEB025; Alisporivir; ribavirin therapy; genotype 2/3 treatment naive patients
MeSH Terms: conditions — Hepatitis C; Liver Diseases; Hepatitis C, Chronic | interventions — alisporivir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 200 mg BID (Experimental): Dual-therapy with a response-guided treatment duration with Alisporivir 200 mg twice daily (BID) and Ribavirin (RBV) for 12 or 24 weeks (Treatment period 1). Patients who were considered treatment failures were to be treated with peg-IFNα2a/RBV 800 mg daily for 24 weeks in Treatment period 2 (Roll-over treatment arm).
  Interventions: Drug: Alisporivir; Drug: Ribavirin; Drug: Peg-IFNα2a
- 300 mg BID (Experimental): Dual-therapy with a response-guided treatment duration with Alisporivir 300mg BID and RBV for 12 or 24 weeks (Treatment period 1). Patients who were considered treatment failures were to be treated with peg-IFNα2a/RBV 800 mg daily for 24 weeks in Treatment period 2 (Roll-over treatment arm).
  Interventions: Drug: Alisporivir; Drug: Ribavirin; Drug: Peg-IFNα2a
- 400 mg BID (Experimental): Dual-therapy with a response-guided treatment duration with Alisporivir 400 mg BID and RBV for 12 or 24 weeks (Treatment period 1). Patients who were considered treatment failures were to be treated with peg-IFNα2a/RBV 800 mg daily for 24 weeks in Treatment period 2 (Roll-over treatment arm).
  Interventions: Drug: Alisporivir; Drug: Ribavirin; Drug: Peg-IFNα2a

INTERVENTIONS:
Drug: Alisporivir — Alisporivir 100 mg or 200 mg soft gel capsules (SGC) in blister packs for oral administration
  Other Names: DEB025
Drug: Ribavirin — Ribavirin tablets of various strengths for oral administration
  Other Names: RBV
Drug: Peg-IFNα2a — Peg-IFNα2a solution for subcutaneous injection

SUMMARY:
This study will explore the relationship of different DEB025 doses in combination with RBV to pharmacokinetic, pharmacodynamic (i.e. viral load reduction) and safety profiles in chronic hepatitis C GT 2 and 3 treatment naïve patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. No previous treatment for Hepatitis C (HCV) infection (i.e. HCV treatment-naïve)
3. Chronic hepatitis C (G2 or G3) virus infection diagnosed

Exclusion criteria:

1. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of that medication before enrollment.
2. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes
3. Hepatitis B Surface Antigen (HBsAg) positive
4. Human immunodeficiency virus (HIV) positive.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Viral load drop from baseline through Week 12 | Baseline through Week 12
Percentage of participants who developed confirmed Stage II or greater hypertension (SBP ≥ 160 mmHg or DBP ≥ 100 mmHg | within 12 weeks
Change in platelet count from baseline through Week 12. | Baseline through Week 12

SECONDARY OUTCOMES:
Number of participants with Sustained Virologic Response at Week 12 follow-up (SVR12) | 12 weeks after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- Germany (10):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Würzburg
- Poland (3):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
- Sweden (6):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Umeå
- United Kingdom (3):
  - Novartis Investigative Site, Frimley, Surrey
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, London